CLINICAL TRIAL: NCT07265895
Title: Inherited Retinal Diseases: Natural History and Genotype-Phenotype Correlations, Monocentric Retrospective Observational Study
Brief Title: Inherited Retinal Diseases: Natural History and Genotype-Phenotype Correlations
Acronym: IRDs-OSR
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Maurizio Battaglia Parodi, Associate Professor, IRCCS San Raffaele
Other Study IDs: IRDs-OSR
Record Dates: First submitted 2025-11-18; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Retinal Degenerations; Retinitis Pigmentosa (RP); Stargardt Disease
MeSH Terms: conditions — Retinal Degeneration; Retinitis Pigmentosa; Stargardt Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intervention: Observational Cohort — no intervention, natural history study

SUMMARY:
Inherited Retinal Diseases (IRDs) are a heterogeneous group of genetically based degenerative retinal disorders, representing a major cause of visual impairment and blindness in working-age adults. Despite the approval of the first gene therapy for RPE65-related IRD (voretigene neparvovec) in 2017, most IRDs remain untreatable, though many gene therapies are in development. Effective trial design and therapy development require a deep understanding of disease natural history and genotype-phenotype correlations. Over 270 IRD-associated genes are known (e.g., ABCA4, USH2A, RPGR, PRPH2, BEST1), each linked to distinct phenotypes and clinical progression. This retrospective study analyzes clinical, functional, and imaging data (Optical Coherence Tomography, Fundus Autofluorescence, Microperimetry) from a large, genetically characterized IRD cohort at the IRCCS Ospedale San Raffaele up to December 31, 2025. The aims are to describe natural history, define genotype-phenotype relationships, and identify structural and functional outcome measures useful for future clinical trial endpoints, supporting personalized prognosis and trial design.

ELIGIBILITY:
Inclusion Criteria:

1. Participant completed at least one ophthalmological and retinal imaging examination at our center.
2. Clinically diagnosed with IRD, as per familiy history, clinical signs or symptoms, retinal imaging findings.
3. Definitive genetic diagnosis of IRD with adequate molecular test

Exclusion Criteria:

1. Affected by other retinal or optic nerve conditions potentially affecting analyses (diabetic retinopathy, glaucoma).
2. History of retinotoxic medications (i.e., hydroxychloroquine, pentosan polysulfate sodium, tamoxifen, ritonavir, didanosine, MEK inhibitors) intake.
3. Unclear genetic diagnosis.
4. Incomplete or inadequate ophthalmological and imaging tests.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients affected by IRDs genetically confirmed
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Best-corrected Visual Acuity | through study completion, an average of 1 year
  Measured on measured Early Treatment Diabetic Retinopathy Study (ETDRS) charts and recorded in logMAR units
Macular threshold sensitivity | through study completion, an average of 1 year
  Measured in decibels using fundus- tracked MP (e.g., MAIA device) across a standard grid of 68 central loci under standardized mesopic conditions.
  Sensitivity deviation from age-matched normative values will also be computed
Total Macular volume | through study completion, an average of 1 year
  Measured in mm3 on OCT scans
Centra Subfield Thickness | through study completion, an average of 1 year
  Measured in micron on OCT scans
Preserved Ellipsoid zone area | through study completion, an average of 1 year
  Measured in mm2 on OCT scans
Foveal Outer Nuclear Layer thickness | through study completion, an average of 1 year
  Measured in microns on OCT scans
Ellipsoid zone loss area | through study completion, an average of 1 year
  Measured in mm2 on OCT scans
Hyperautofluorescent (Robson- Holder) ring area | through study completion, an average of 1 year
  Measured in mm2 on FAF images
Dereased Autofluorescence area | through study completion, an average of 1 year
  Measured in mm2 on Fundus autofluorescence images

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: No
single center study